CLINICAL TRIAL: NCT00872014
Title: Phase 2 Open-label Multi-Center Study to Evaluate the Efficacy and Safety of AMG 386 and Sorafenib as First Line Therapy for Subjects With Advanced or Inoperable Hepatocellular Carcinoma
Brief Title: A Study of the Effectiveness and Safety of AMG 386 and Sorafenib to Treat Advanced or Inoperable Hepatocellular Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080580
Record Dates: First submitted 2009-03-12; First posted 2009-03-30 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-02

CONDITIONS: Advanced Hepatocellular Carcinoma; Inoperable Hepatocellular Carcinoma
MeSH Terms: interventions — trebananib; Sorafenib

ARMS (2):
- 15mg/ kg cohort (Experimental): AMG 386 15mg/kg intravenously once weekly and Sorafenib 400mg orally twice daily in an every 4 weeks dosing schedule.
  Interventions: Drug: AMG 386; Drug: Sorafenib
- 10 mg/kg cohort (Experimental): AMG 386 10mg/kg intravenously once weekly and Sorafenib 400mg orally twice daily in an every 4 weeks dosing schedule.
  Interventions: Drug: AMG 386; Drug: Sorafenib

INTERVENTIONS:
Drug: AMG 386 — Two doses of AMG 386 (15 mg/kg) IV QW will be studied
  Arms: 15mg/ kg cohort
Drug: AMG 386 — Two doses of AMG 386 (10 mg/kg) IV QW will be studied
  Arms: 10 mg/kg cohort
Drug: Sorafenib — Sorafenib 400 mg PO BID orally twice daily in an every 4 week dosing schedule for 15mg/kg cohort & 10mg/kg cohort

SUMMARY:
The purpose of this study is to determine whether AMG 386, in combination with Sorafenib, is effective in the treatment of advanced or inoperable Hepatocellular cancer in subjects who have not received any prior systemic therapy except surgery or locoregional therapy.

Disease status and disease progression will be assessed every 8 weeks. Subjects will remain on treatment until: progressive disease by RECIST criteria; clinical progression; death or loss to follow-up; or withdrawal of informed consent.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of AMG 386 in combination with sorafenib as measured by the progression free survival (PFS) rate at 4 months in subjects with advanced or inoperable hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or inoperable HCC
* Child-Pugh A liver function score
* Measurable disease with at least one unidimensionally measurable lesion per RECIST 1.0 guidelines with modifications
* Adequate organ and hematological function
* Men or women greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less

Exclusion Criteria:

* Subject is eligible for a liver transplant per investigators discretion
* Any previous systemic chemotherapy for HCC
* History of arterial or venous thromboembolism within 12 months prior to enrollment
* History of clinically significant bleeding within 6 months prior to enrollment
* History of central nervous system metastases
* Clinically significant cardiovascular disease within 12 months
* Uncontrolled hypertension
* Subjects with a history of prior malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) rate at 4 months | 4 months

SECONDARY OUTCOMES:
Incidence of adverse events and significant laboratory abnormalities | Adverse events at every visit, significant laboratory abnormalities at least every 4 weeks
Objective response rate, Disease control rate, Progression free survival, Overall survival, Time to progression | Radiologic imaging every 8 weeks
Pharmacokinetic parameters for AMG 386 when used in combination with Sorafenib | Weeks 1, 2, 5, 9, and every 16 weeks thereafter
Pharmacokinetic parameter for Sorafenib when used in combination with AMG 386 | Weeks 2, 5, 9, and every 16 weeks thereafter
Incidence of the occurrence of anti-AMG 386 antibody formation | Weeks 1, 5, 9, and every 16 weeks thereafter
Baseline values of and changes from baseline in pharmacodynamic, immunologic, biochemical, transcriptional, pharmacogenetic and angiogenic markers | Weeks 1, 2, 5, and every 16 weeks thereafter

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Abou-Alfa GK, Blanc JF, Miles S, Ganten T, Trojan J, Cebon J, Liem AK, Lipton L, Gupta C, Wu B, Bass M, Hollywood E, Ma J, Bradley M, Litten J, Saltz LB. Phase II Study of First-Line Trebananib Plus Sorafenib in Patients with Advanced Hepatocellular Carcinoma. Oncologist. 2017 Jul;22(7):780-e65. doi: 10.1634/theoncologist.2017-0058. Epub 2017 Jun 7. PMID 28592620
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com